CLINICAL TRIAL: NCT01429688
Title: A Randomized, Single-dose, 2-sequence, 2-period Crossover Study to Investigate the Food-effect Pharmacokinetics of Sarpogrelate HCl Controlled Release Tablet in Healthy Male Subjects
Brief Title: Pharmacokinetic / Pharmacodynamic (PK/PD) Study of Multiple Doses of DP-R202 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DP-SACL-I-003
Record Dates: First submitted 2011-08-29; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP-R202 (Experimental): Multiple oral administration for 3 days
  Interventions: Drug: Anplag
- Anplag (Active Comparator): Multiple oral administration for 3days
  Interventions: Drug: Anplag

INTERVENTIONS:
Drug: Anplag — Sarpogrelate HCl 300mg once a day or 100mg three times a day for 3 days
  Other Names: Other Names:; DP-R202 : DP11002-3; Anplag : 0007-1

SUMMARY:
The purpose of this study is compare the safety and pharmacokinetic characteristics of DP-R202 (Sarpogrelate HCl 100mg, qd) with those of Anplag (Sarpogrelate HCl 100mg, tid) after multiple oral administration in healthy male volunteers.

DETAILED DESCRIPTION:
The number of patient is thirthy-six.Patients were randomly assigned either anplag tablet(Sarpogrelate HCL 100mg, tid)3days first, DP-R202(Sarpogrelate HCL 300mg, qd) 3days Second or DP-R202(Sarpogrelate HCL 300mg, qd)3days first, anplag tablet(Sarpogrelate HCL 100mg, tid) 3days second.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Sarpogrelate HCL or other antiplatelets

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics | comparator 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 6.33, 6.67, 7, 7.5, 8, 9, 12, 12.33, 12.67, 13, 13.5, 14, 15, 16, 24h Test drug : 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24h
  Cmax, ss, AUCτ

SECONDARY OUTCOMES:
Composite of pharmacokinetics | comparator 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 6.33, 6.67, 7, 7.5, 8, 9, 12, 12.33, 12.67, 13, 13.5, 14, 15, 16, 24h Test drug : 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24h
  tmax,ss, t1/2, Cav,ss, PTF, AI, Cmin,ss

CONTACTS AND LOCATIONS:
Overall Officials: Jae Wook Ko, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea